CLINICAL TRIAL: NCT07238504
Title: Acupuncture for Post-hemorrhoidectomy Pain Control With Acute Anti-inflammatory Effects: A Randomized Controlled Trial
Brief Title: Acupuncture for Post-hemorrhoidectomy Pain Control
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: School of Chinese Medicine, The University of Hong Kong (Unknown)
Responsible Party: Principal Investigator, Pak Chiu WONG, Associate Consultant, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 25-302
Record Dates: First submitted 2025-09-24; First posted 2025-11-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hemorrhoidectomy; Hemorrhoid Pain; Acupuncture
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fully active acupuncture (Experimental)
  Interventions: Procedure: Acupuncture
- Minimum acupuncture stimulation (Sham Comparator)
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture to 6 specific acupoints, 3 distant acupoints and electrical stimulation to 4 pairs of local acupoints.
  Other Names: Fully active acupuncture
  Arms: Fully active acupuncture
Procedure: Acupuncture — Minimal electrical stimulation to 1 local acupoint and 2 distant acupoints
  Other Names: Minimum acupuncture stimulation
  Arms: Minimum acupuncture stimulation

SUMMARY:
The goal of this clinical trial is to learn if acupuncture improves pain control after hemorrhoidectomy in patients with symptomatic hemorrhoids. It will also learn about the safety of using acupuncture in surgical patients. The main questions it aims to answer are:

Does acupuncture lower the maximal pain intensity after hemorrhoidectomy? Does acupuncture reduce analgesics requirement, length of hospital stay and quality of recovery?

Researchers will compare fully active acupuncture to a sham treatment (a look-alike procedure with minimum acupuncture stimulation) to see if active acupuncture works to improve pain control.

Participants will:

Receive acupuncture treatment for 7 times over first 5 days after surgery. Visit the clinic once 2 weeks after surgery for checkups and tests. Keep a diary of their symptoms and the number of times they take pain-killers.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic grade III or IV hemorrhoids undergoing conventional hemorrhoidectomy

Exclusion Criteria:

1. Patients scheduled for stapled hemorrhoidopexy
2. Concomitant surgery other than conventional hemorrhoidectomy
3. Bleeding tendency, thrombocytopenia (platelet count < 100 x 10^9/L)
4. Immunocompromised status or use of chemotherapy
5. Active dermatitis
6. Patients with pacemaker or automated implantable cardioverter-defibrillator
7. Pregnant patients
8. Known allergy to opioids, local anaesthetic drugs, paracetamol, non-steroidal anti-inflammatory drugs (NSAIDS) including cyclooxygenase-2 inhibitors
9. History of chronic pain (duration for 3 months or more)
10. Daily use of strong opioids (e.g. morphine, fentanyl, hydromorphone, methadone, oxycodone, or meperidine)
11. Alcohol or drug abuse
12. Psychiatric illness
13. Impaired renal function (preoperative serum creatinine level > 120µmol/L)
14. Recent acupuncture treatment for other medical conditions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Maximal pain intensity | Post-operative day 1
  Numeric rating scale (minimum at 0 means 'no pain', maximum at 10 means 'worst pain')

SECONDARY OUTCOMES:
Maximal and resting pain intensity | Post-operative day 0, 2 to 7 and 14
  Numeric rating scale (minimum at 0 means 'no pain', maximum at 10 mean 'worst pain')
Dosage of analgesics requirement | Post-operative 2 weeks
  Dosage of paracetamol, tramadol and celecoxib tablets taken per day over the first post-operative 2 weeks
Length of hospital stay | Post-operative day 1
Functional recovery questionnaire | Post-operative 1 week (time to first bowel motion, time to first urination and time to return to work, counted from the day of operation)
Adverse effect | Post-operative 2 weeks
  Effect from analgesics and acupuncture
Quality of recovery (QoR) | Post-operative day 1
  QoR-15 questionnaire, which includes 15 questions scoring at a 10-point scale. Minimum at 0 means worst outcome and maximum at 10 means best outcome.
Serum C-reactive protein level | Post-operative day 0 and 1

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT07238504/Prot_SAP_ICF_000.pdf